CLINICAL TRIAL: NCT00882440
Title: A Double-Blind, Randomized, Parallel, Placebo-Controlled Study to Investigate the Antihypertensive Efficacy and Safety of Different Doses of DuP 753 (MK0954)
Brief Title: A Study to Investigate the Efficacy and Safety of Different Doses of Losartan Potassium (MK0954-011)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0954-011; MK0954-011; 2009_574
Record Dates: First submitted 2009-04-14; First posted 2009-04-16 (Estimated); Results first posted 2009-06-10 (Estimated); Last update posted 2015-08-27 (Estimated); Status verified 2015-08

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension | interventions — Losartan; Enalapril

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (7):
- 1 (Placebo Comparator): Placebo
  Interventions: Drug: Placebo
- 2 (Experimental): Losartan 10 mg
  Interventions: Drug: losartan potassium
- 3 (Experimental): Losartan 25 mg
  Interventions: Drug: losartan potassium
- 4 (Experimental): Losartan 50 mg
  Interventions: Drug: losartan potassium
- 5 (Experimental): Losartan 100 mg
  Interventions: Drug: losartan potassium
- 6 (Experimental): Losartan 150 mg
  Interventions: Drug: losartan potassium
- 7 (Active Comparator): Enalapril 20 mg
  Interventions: Drug: Enalapril

INTERVENTIONS:
Drug: losartan potassium — losartan oral capsule (10, 25, 50, 100 or 150 mg) once daily for 8 weeks
  Other Names: MK0954; Cozaar
  Arms: 2; 3; 4; 5; 6
Drug: Placebo — Placebo capsule to losartan
  Arms: 1
Drug: Enalapril — Enalapril 20 mg oral tablet taken once daily for 8 weeks
  Arms: 7

SUMMARY:
The purpose of this study was to compare the antihypertensive efficacy of different doses of losartan compared to placebo and enalapril, in patients with supine diastolic blood pressure of 100-115 mmHg.

ELIGIBILITY:
Inclusion Criteria:

* Patient has been diagnosed with mild to moderate hypertension, with supine diastolic blood pressure of 100 to 115 mmHg
* Patient has no active medical problems other than essential hypertension that might affect blood pressure
* Patient has received no drug therapy that might affect blood pressure

Exclusion Criteria:

* Prior exposure to losartan
* History of stroke
* History of myocardial infarction
* Atrial flutter or atrial fibrillation
* History of congestive Heart failure
* Known Sensitivity to ACE inhibitors
* Known positive test for HIV/AIDS or Hepatitis B
* Patient is being treated for acute ulcer disease
* History of chronic liver disease
* Actively treated diabetes mellitis
* Any known bleeding or platelet disorder
* Absence of one kidney
* Women of childbearing potential or who are breastfeeding
* Patient is abusing or has a history of alcoholism or drug addiction

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 576 (Actual)
Dates: Start 1990-12; Primary Completion 1991-08 (Actual); Study Completion 1992-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Background] Gradman AH, Arcuri KE, Goldberg AI, Ikeda LS, Nelson EB, Snavely DB, Sweet CS. A randomized, placebo-controlled, double-blind, parallel study of various doses of losartan potassium compared with enalapril maleate in patients with essential hypertension. Hypertension. 1995 Jun;25(6):1345-50. doi: 10.1161/01.hyp.25.6.1345. PMID 7768585

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited at 28 sites in the United States. Primary Therapy Period: December, 1990-August, 1991
Pre-assignment Details: Patients could be randomized after the 4-week placebo baseline period if their mean supine diastolic blood pressure (SuDBP) was 100-115 mmHg and ≤7 mmHg from the mean SuDBP after 2 weeks of placebo therapy, or after a 2-week placebo baseline period if 2 sets of SuDBP data were within 100-115 mmHg, ≥3 days apart and differed by ≤7 mmHg.
Groups:
- Placebo: Losartan and Enalapril placebo orally once daily for 8 weeks
- Losartan 10 mg: Losartan 10 mg orally once daily for 8 weeks
- Losartan 25 mg: Losartan 25 mg orally once daily for 8 weeks
- Losartan 50 mg: Losartan 50 mg orally once daily for 8 weeks
- Losartan 100 mg: Losartan 100 mg orally once daily for 8 weeks
- Losartan 150 mg: Losartan 150 mg orally once daily for 8 weeks
- Enalapril 20: Enalapril 20 mg orally once daily for 8 weeks
Period: Overall Study
Arm/Group | Placebo | Losartan 10 mg | Losartan 25 mg | Losartan 50 mg | Losartan 100 mg | Losartan 150 mg | Enalapril 20
Started | 78 | 80 | 82 | 79 | 90 | 84 | 83
Completed | 67 | 72 | 75 | 76 | 80 | 77 | 79
Not Completed | 11 | 8 | 7 | 3 | 10 | 7 | 4
Not completed — Adverse Event | 2 | 2 | 2 | 1 | 1 | 4 | 2
Not completed — Lack of Efficacy | 3 | 5 | 2 | 0 | 0 | 3 | 0
Not completed — Lost to Follow-up | 2 | 0 | 1 | 1 | 1 | 0 | 1
Not completed — Protocol Violation | 0 | 0 | 1 | 1 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 2 | 1 | 1 | 0 | 6 | 0 | 1
Not completed — Patient Uncooperative | 2 | 0 | 0 | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Losartan 10 mg | Losartan 25 mg | Losartan 50 mg | Losartan 100 mg | Losartan 150 mg | Enalapril 20 | Total
Number analyzed (Participants) | 78 | 80 | 82 | 79 | 90 | 84 | 83 | 576
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.3 (11.6) | 53.9 (12.3) | 52.8 (12.2) | 52.8 (10.3) | 54.0 (10.2) | 53.9 (10.8) | 51.9 (11.1) | 53.1 (11.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31 | 29 | 27 | 26 | 31 | 22 | 27 | 193
  Male | 47 | 51 | 55 | 53 | 59 | 62 | 56 | 383
Race/Ethnicity [Number; unit: participants]
  Caucasian | 64 | 60 | 63 | 57 | 66 | 64 | 64 | 438
  Black | 5 | 10 | 14 | 11 | 17 | 11 | 7 | 75
  Hispanic | 9 | 9 | 5 | 11 | 7 | 8 | 10 | 59
  Other | 0 | 1 | 0 | 0 | 0 | 1 | 2 | 4
SuDBP [Mean (Standard Deviation); unit: mmHg] — Supine Diastolic Blood Pressure (SuDBP)
  mmHg | 103.3 (3.8) | 104.3 (3.9) | 103.3 (3.7) | 104.0 (3.7) | 104.1 (4.2) | 103.4 (3.4) | 103.1 (3.7) | 103.7 (3.8)

OUTCOME MEASURES:

1. Secondary Outcome: Categories of Antihypertensive Response in Trough Supine Diastolic Blood Pressure (SuDBP) at Week 8
Description: Patients in Category I (defined as "excellent" in protocol) if SuDBP was <90 mmHg, Category II (defined as "good" in protocol) if SuDBP was ≥90 but decreased at least 10 mmHg, or Category III (defined as "fair" or "inadequate" in protocol) if SuDBP was ≥90 and decreased less than 10 mmHg.
Time Frame: 24 hours post dose at Week 8
Population: An "all patients treated" approach was employed that included patients with at least one treatment period measurement. The last measurements of withdrawn patients were carried forward to subsequent timepoints. Missing data were estimated by carrying forward data from the last visit (excluding baseline) at which it was available.
Measure: Number; unit: Participants
Arm/Group | Placebo | Losartan 10 mg | Losartan 25 mg | Losartan 50 mg | Losartan 100 mg | Losartan 150 mg | Enalapril 20
Number analyzed (Participants) | 78 | 80 | 82 | 78 | 89 | 84 | 82
Participants
  Category I | 10 | 19 | 21 | 24 | 29 | 28 | 35
  Category II | 14 | 17 | 7 | 15 | 19 | 12 | 16
  Category III | 54 | 44 | 54 | 39 | 41 | 44 | 31

2. Primary Outcome: Mean Change From Baseline in Trough Supine Diastolic Blood Pressure (SuDBP) at Week 8
Time Frame: 24 hours post dose at Baseline and Week 8
Population: The primary analysis employed an "all patients treated" approach that included patients with at least one treatment period measurement. The last measurements of withdrawn patients were carried forward to subsequent timepoints. Missing data were estimated by carrying forward data from the last visit (excluding baseline) at which it was available.
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Placebo | Losartan 10 mg | Losartan 25 mg | Losartan 50 mg | Losartan 100 mg | Losartan 150 mg | Enalapril 20
Number analyzed (Participants) | 78 | 80 | 82 | 78 | 89 | 84 | 82
mm Hg | -5.6 (7.8) | -7.9 (7.6) | -6.8 (7.9) | -10.1 (7.0) | -9.9 (6.9) | -9.7 (8.0) | -11.2 (6.7)

3. Secondary Outcome: Mean Change From Baseline in Peak Supine Diastolic Blood Pressure (SuDBP) at Week 8
Time Frame: 6 hours post dose at Baseline and 8 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Placebo | Losartan 10 mg | Losartan 25 mg | Losartan 50 mg | Losartan 100 mg | Losartan 150 mg | Enalapril 20
Number analyzed (Participants) | 75 | 79 | 80 | 77 | 87 | 81 | 82
mm Hg | -4.7 (8.7) | -7.3 (9.4) | -9.9 (8.5) | -11.9 (9.2) | -10.4 (8.9) | -13.1 (9.0) | -16.2 (10.4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Merck agreements may vary with individual investigators, but will not prohibit any investigator from publishing. Merck supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.